CLINICAL TRIAL: NCT01831752
Title: Performance Evaluation of a Non-Invasive Glucose Monitor (Spectral Data Acquisition) as Compared to CGM Data Acquired by the iPro2
Brief Title: Performance Evaluation of a Non-Invasive Glucose Monitor as Compared to CGM Data Acquired by the iPro2
Status: Completed | Type: Observational
Sponsor: Sansum Diabetes Research Institute (Other)
Responsible Party: Principal Investigator, Kristin Castorino, DO, Principal Investigator, Sansum Diabetes Research Institute
Other Study IDs: ZY001
Record Dates: First submitted 2013-03-05; First posted 2013-04-15 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes; Type 1; Continuous glucose monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 1 Diabetes Melitus: Subjects aged 12 through 75, previously diagnosed with type 1 diabetes mellitus, currently using insulin to treat their diabetes.

SUMMARY:
This study is for adults and adolescents with type 1 diabetes. The purpose of this study is to learn more about an investigational system to measure blood glucose. This system does not require blood to be drawn from the body, and it does not require a glucose sensor to be worn under the skin (subcutaneously). This device instead estimates blood glucose levels by shining infrared light on the skin and then using sophisticated statistical analysis on how the light bounces back or gets absorbed (spectral data). The researchers in this study will compare the accuracy of the new device to glucose measurement devices that are already approved by the FDA, including glucose meters and subcutaneous continuous glucose monitoring (CGM) sensors. Information learned from this study will be used in the development of tools for managing diabetes.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the utility of a novel approach to non-invasive glucose sensing. The testing for each patient includes fingerstick and alternate site capillary blood measurements taken nearly simultaneously with a series of near-infrared spectra collected via a novel, proprietary fiber-optic probe. Simultaneously, subjects will be wearing a commercial continuous glucose measuring system (Medtronic iPro 2). The spectral data are converted to a prediction of tissue glucose using a proprietary pre-defined universal algorithm. Subjects are tested every 20 minutes for up to 12 hours per day and up to 6 visits per patient over a period of up to 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 12-75 years
* Have been diagnosed with type 1 diabetes mellitus
* Use insulin to treat your diabetes
* Agree and are able to follow the study plans as described in this informed consent form.

Exclusion Criteria:

* Are a pregnant woman or nursing mother
* Have skin conditions that could cause a problem wearing a glucose sensor on your abdomen (stomach area) and/or having spectral data measured from your forearm with the non-invasive device.
* Are currently taking part in another clinical study
* Have taken part in this study before
* Have experienced severe hypoglycemia (an episode of low blood sugar that you were unable to treat yourself - e.g., seizure, coma, unconsciousness) any time within the past six months
* Have any additional condition(s) that in the Investigator's opinion would warrant exclusion from the study or prevent you from completing the study

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects aged 12 through 75, previously diagnosed with type 1 diabetes mellitus, currently using insulin to treat their diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2013-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
blood glucose correlation coefficient | Up to 16 weeks
  To generate a non-invasive blood glucose measurement with continuous glucose monitor data and alternate site data.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Zisser, MD, Principal Investigator — Sansum Diabetes Research Institute
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States